CLINICAL TRIAL: NCT01574014
Title: Glucocorticoid Treatment for Social Phobia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruiting problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161/07; 32003B_124947 (Other Grant/Funding Number: SNF); 2008DR2002 (Other: Swissmedic)
Record Dates: First submitted 2012-03-14; First posted 2012-04-10 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Phobic Disorders; Phobias
Keywords: Anxiety Disorder; Phobic Disorders
MeSH Terms: conditions — Phobic Disorders; Anxiety Disorders | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: CBGT & Hydrocortisone (Active Comparator)
  Interventions: Behavioral: CBGT; Drug: Hydrocortisone
- 2: CBGT & Placebo (Placebo Comparator)
  Interventions: Behavioral: CBGT; Drug: Placebo

INTERVENTIONS:
Behavioral: CBGT — Cognitive-behavioral group therapy
Drug: Hydrocortisone — 3 x 20 mg Hydrocortisone (oral, 60 min. before MRI1, 60 min. before exposition in CBGT1 and 60 min. before exposition in CBGT2)
  Arms: 1: CBGT & Hydrocortisone
Drug: Placebo — Placebo (oral, 60 min. before MRI1, 60 min. before exposition in CBGT1 and 60 min. before exposition in CBGT2)
  Arms: 2: CBGT & Placebo

SUMMARY:
Social phobia is the third most common psychiatric disorder besides depression and alcoholism. Several studies have demonstrated the efficacy of cognitive-behavioral therapy in the treatment of social phobia. Nevertheless, there is no effect in a third of the people at the existing treatment methods. Pharmacological therapies have similar effects, but there is a high rate of relapse after discontinuation of medication.

Social phobia is characterized by fear of performance or interaction situations. The strong fear of negative evaluation by others is usually accompanied by a marked avoidance behavior and increased physical symptoms such as blushing, sweating, palpitations, or tremors. The confrontation with a phobic stimulus leads to a retrieval of stimulus-associated aversive memories, resulting in an immediate anxiety response. Several studies had already shown that elevated glucocorticoids impair retrieval of declarative memory contents in healthy subjects. The investigators demonstrated an anxiety-reducing effect after the administration of cortisone before the confrontation with a phobic stimulus in patients with social and spider phobia.

DETAILED DESCRIPTION:
Background

Anxiety disorders have major public health significance and social phobia ranks as the third most common mental health disorder after depression and alcoholism. Even though cognitive-behavioral therapy (CBT) is the most effective non-pharmacological approach to the treatment of social phobia, more than one third of the patients do not respond to treatment, or achieve only partial remission of symptoms. Pharmacotherapy (e.g., SSRIs, benzodiazepines) has been shown to be effective in the acute treatment of social phobia, however, with high rates of relapse when medication is discontinued. In addition, the combination of CBT and medication does not seem to be more beneficial than CBT alone. Consequently, the development of innovative psychobiological approaches combining effective psychotherapy methods with synergizing substance administration is a primary challenge in interdisciplinary research on treatment of social phobia.

In a recent study the investigators found evidence that a pharmacological elevation of glucocorticoid levels reduces fear in patients with social phobia and spider phobia exposed to a phobic stimulus. Furthermore, the investigators have shown that repeated administration of glucocorticoids before exposure to a phobic stimulus leads to an extinction of phobic fear. Also the low-dose administration of cortisone over a month in patients with post-traumatic stress disorder reduces cardinal of symptoms the disorder. Based on these findings, glucocorticoid treatment, in combination with exposure therapy, may help to reduce fear and promote extinction of phobic fear.

In an interdisciplinary research project involving psychology, behavioral pharmacology psychiatry, genetics and neuroimaging the investigators propose to investigate the therapeutic efficacy of combining an exposure-based cognitive-behavioral group therapy (CBGT) with hydrocortisone treatment. The investigators hypothesize that hydrocortisone exerts both acute beneficial effects by reducing fear during exposure, and long-term beneficial effects by facilitating the extinction of phobic fear. Furthermore, the investigators hypothesize differential treatment responses depending on genetic variations in glucocorticoid-related genes (substudy 1). These hypotheses will be tested in a clinical study with 100 patients with mainly speech anxiety who fulfill DSM-IV criteria for a diagnosis of social phobia and 60 patients with spider phobia.

This is the first study aimed at determining the therapeutic efficacy of combining hydrocortisone administration and a short-term exposure-based cognitive-behavioral group therapy for the treatment of social phobic patients with specific speech anxiety and patients with spider phobia. Considering the large number of patients suffering from social phobia, the suggested interdisciplinary project will have important clinical implications for the development of a more effective therapy.

Objective

To determine whether short-term treatment with 20 mg hydrocortisone enhances the efficacy of exposure-based cognitive-behavioral group therapy (CBGT) in patients with social phobia, specifically speech anxiety and patients with spider phobia.

A series of studies indicate that elevated glucocorticoid levels inhibit the retrieval of memory in healthy humans. Further the low-dose administration of glucocorticoids over a month inhibited the retrieval of traumatic memories in patients with post traumatic stress disorder. These findings suggest that glucocorticoids might also inhibit retrieval of fear memory in phobia and social phobia exposed to a phobic stimulus. Additionally, the investigators found evidence indicating that repeated administration of glucocorticoids before exposure to a phobic stimulus leads to an extinction of phobic fear. Based on these findings, glucocorticoid treatment, in combination with exposure therapy, may help to reduce fear and promote extinction of phobic fear.

Methods

In a placebo-controlled double-blind study design, patients will be randomly assigned to receive CBGT + hydrocortisone (Social Phobia: N=50 / Spider Phobia: N=30) or CBGT + placebo (Social Phobia: N=50 / Spider Phobia: N=30). Psychopathological symptoms and stress reactivity will be assessed by psychometric and endocrine parameters before, during and after CBGT therapy. The patients have further the possibility to attend to a neuroimaging study, in which the investigators examine and localize the anxiolytic effect of acute glucocorticoid administration in the brain (substudy 2). In this substudy 2 the investigators compare the patients with social phobia with patients with specific spider phobia and healthy controls as they did in their previous studies (Soravia et al. 2006).

ELIGIBILITY:
Inclusion Criteria:

* Age (20-55)
* Spider Phobia
* Right Handed
* Social Phobia

Exclusion Criteria:

* Other Psychiatric Disorder / Comorbidities
* Smoking more than 15 cigarettes per day
* Medication
* Contraceptives
* Physical illness
* Neurological disease
* Drug abuse

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2009-07; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in spider phobia symptoms / social phobia symptoms | at follow-up visit, expected to be after 3 months
  measured by various standardized questionnaires

SECONDARY OUTCOMES:
Change from baseline in state and trait anxiety | 1-3 weeks before treatment, 4 weeks after treatment, 3 months after treatment
  measured by standardized questionnaires
Change from baseline in personality traits | 1-3 weeks before treatment
  measured by standardized questionnaires
Change from baseline in amygdala activation | 1-3 weeks before treatment, 4 weeks after treatment
  measured by several magnetic resonance sequences

CONTACTS AND LOCATIONS:
Overall Officials: Leila M Soravia, PhD, Principal Investigator — Department of Psychiatric Neurophysiology, University Hospital of Psychiatry, University of Bern
Locations (1):
- Dep. of Psychiatric Neurophysiology, University Hospital of Psychiatry, University of Bern, Bern, Switzerland

REFERENCES:
- [Background] Soravia LM, de Quervain DJ, Heinrichs M. Glucocorticoids do not reduce subjective fear in healthy subjects exposed to social stress. Biol Psychol. 2009 Jul;81(3):184-8. doi: 10.1016/j.biopsycho.2009.04.001. Epub 2009 Apr 11. PMID 19482235
- [Background] de Quervain DJ, Roozendaal B, Nitsch RM, McGaugh JL, Hock C. Acute cortisone administration impairs retrieval of long-term declarative memory in humans. Nat Neurosci. 2000 Apr;3(4):313-4. doi: 10.1038/73873. No abstract available. PMID 10725918
- [Background] de Quervain DJ, Roozendaal B, McGaugh JL. Stress and glucocorticoids impair retrieval of long-term spatial memory. Nature. 1998 Aug 20;394(6695):787-90. doi: 10.1038/29542. PMID 9723618
- [Background] Aerni A, Traber R, Hock C, Roozendaal B, Schelling G, Papassotiropoulos A, Nitsch RM, Schnyder U, de Quervain DJ. Low-dose cortisol for symptoms of posttraumatic stress disorder. Am J Psychiatry. 2004 Aug;161(8):1488-90. doi: 10.1176/appi.ajp.161.8.1488. PMID 15285979
- [Derived] Soravia LM, Schwab S, Weber N, Nakataki M, Wiest R, Strik W, Heinrichs M, de Quervain D, Federspiel A. Glucocorticoid administration restores salience network activity in patients with spider phobia. Depress Anxiety. 2018 Oct;35(10):925-934. doi: 10.1002/da.22806. Epub 2018 Aug 12. PMID 30099829